CLINICAL TRIAL: NCT03702036
Title: Compassionate Use Individual Request Program for GSK525762 in NUT Midline Carcinoma
Status: No longer available | Type: Expanded Access
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 209447
Record Dates: First submitted 2018-10-04; First posted 2018-10-10 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Solid Tumours
Keywords: Nuclear protein in testis (NUT); NUT Midline Carcinoma (NMC)
MeSH Terms: interventions — molibresib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: molibresib — molibresib 20 mg will be supplied for compassionate use for the identified individual subject.

SUMMARY:
Compassionate use access to molibresib/GSK525762 for eligible participant with NUT Midline Carcinoma; indication is a seriously debilitating or life-threatening disease.

DETAILED DESCRIPTION:
Investigational Product GSK525762 is an orally bioavailable small molecule that is a potent inhibitor of the binding of BET proteins to acetylated histones. Binding of GSK525762 induces squamous differentiation and inhibits proliferation of patient-derived NMC cell lines both in culture and in murine xenografts.

Compassionate use access to molibresib is restricted to patients with confirmed diagnosis of NUT Midline Carcinoma.

ELIGIBILITY:
Inclusion Criteria

1. Participants meeting all three of the following criteria will be eligible:

   * Diagnosis of NUT Midline Carcinoma based on ectopic expression of NUT protein as determined by IHC and/or detection of NUT gene translocation as determined by FISH.
   * there is no satisfactory alternative treatment; and
   * there is reason to believe that the benefit:risk ratio for molibresib in the indication is positive.
2. Written informed consent can be obtained from the participant or legally authorised representative.
3. Participant must be ≥16 years of age, at the time of signing the informed consent.
4. Demonstrate adequate organ function defined as :Hematological Absolute neutrophil count (ANC) ≥1.5 X 109/liter (L) ; Platelets ≥100 X 109/L ; Hemoglobin≥9.0 g/deciliter ; total bilirubin ≤ 1.5 x X ULN (upper limit of normal)(isolated bilirubin >1.5 X ULN is acceptable if bilirubin is fractionated and direct bilirubin <35% or participant has a diagnosis of Gilbert's syndrome) ; Alanine transaminase ≤ 2.5 X ULN OR ≤ 5 X ULN with documented liver metastases/tumor infiltration; Prothrombin Time (PT) or Partial Thromboplastin Time (PTT) ≤ 1.5 X upper limit of normal (ULN); Renal creatinine OR calculated creatinine clearance [calculated or directly measured] ≤1.5 X ULN or ≥ 50 mL/min; Ejection fraction ≥ Lower limit of normal (LLN); Troponin ≤ ULN
5. Female participants who are not pregnant, breastfeeding and at least one of the following applies:

   a. Is not a woman of childbearing potential (WOCBP) OR Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year, see Appendix 5), preferably with low user dependency, during the intervention period and for at least 7 months after the last dose of molibresib. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of molibresib.
6. Female participants of childbearing potential: Negative highly sensitive serum pregnancy test (as required by local regulations) within 72 hours prior to the first dose of molibresib.
7. NOTE: The investigator is responsible for review of medical history, menstrual history and recent sexual activity to decrease risk for inclusion of a woman with an early undetected pregnancy.
8. Male participants are eligible to participate if agree to the following during intervention period and for at least 16 weeks after the last dose of molibresib:
9. Refrain from donating sperm
10. PLUS, if have a female partner of childbearing potential, either:

Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent -OR- Agree to use a male condom and if female partner is not pregnant, partner to use an additional highly effective contraceptive method with a failure rate of <1% per year.

Exclusion Criteria

1. Use of anticoagulants (e.g., warfarin, heparin) at therapeutic levels within 7 days prior to the first dose of molibresib. Low dose (prophylactic) anticoagulants (e.g., low molecular weight heparin (LMWH) or oral anticoagulants) is permitted. In addition, INR must be monitored in accordance with local institutional practices, as appropriate.
2. Concurrent use of non-steroidal anti-inflammatory drugs (NSAIDs) except for cases where NSAIDs provide benefit over other analgesics or high dose aspirin (allowed up to 100 mg PO daily).
3. Participants with a history of known bleeding disorder(s) or history of clinically significant hemorrhage (e.g., GI, neurologic) within the past 6 months.
4. Evidence of cardiac abnormalities as evidenced by any of the following:

   * History or current clinically significant conduction abnormalities, uncontrolled arrhythmias or hypertension.
   * History or evidence of current ≥Class II congestive heart failure as defined by New York Heart Association (NYHA).
   * Recent history (within the past 3 months) of acute coronary syndromes (including unstable angina and myocardial infarction), coronary angioplasty, or stenting
   * Baseline QTcF interval ≥480 msec
5. Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones, liver metastases or otherwise stable chronic liver disease per investigator assessment).
6. Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, hepatic, renal, cardiac disease, or clinically significant bleeding episodes). Any serious and/or unstable pre-existing medical or psychiatric disorder, or other conditions that could interfere with participant's safety, obtaining informed consent or compliance in the opinion of the investigator.
7. Presence of hepatitis B surface antigen (HBsAg) or positive hepatitis C antibody test result at screening.

   NOTE: Participants with positive Hepatitis C antibody due to prior resolved disease can be enrolled only if a confirmatory negative Hepatitis C RNA PCR is obtained.
8. History of known HIV infection.
9. Hemoptysis >1 teaspoon in 24 hours within the last 28 days.
10. GSK525762 is a benzodiazepine class molecule. Any serious known immediate or delayed hypersensitivity reaction(s) to molibresib or idiosyncrasy to drugs chemically related to molibresib.

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline